CLINICAL TRIAL: NCT01737424
Title: A Dose Blocked-randomized, Double-blind, Placebo-controlled, Single Dosing and Dose-escalation Phase I Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetic Characteristics of LC28-0126 in Healthy Male Subjects
Brief Title: Study to Investigate the Safety and Pharmacokinetic Characteristics of LC28-0126 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-CYCL001
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- LC28-0126 (Experimental): LC28-0126(IV)
  Interventions: Drug: LC28-0126

INTERVENTIONS:
Drug: LC28-0126 — LC28-0126
  Arms: LC28-0126
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To investigate the safety, tolerability and pharmacokinetic characteristics of LC28-0126 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 20 and 45 years at screening.
* Subjects with BMI between 18.0(inclusive) and 27.0 kg/m2 (exclusive); and a total body weight between 55 kg (inclusive) and 90 kg (exclusive)

Exclusion Criteria:

* Participation in a clinical research study within the previous 2 months
* Regular alcohol consumption >21 units per week.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Adverse events | 12 days

SECONDARY OUTCOMES:
Cmax | up to 6 days post-dose
AUC | up to 6 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea